CLINICAL TRIAL: NCT05649475
Title: Circulating Tumor DNA Monitoring in Breast Cancer Undergoing Neoadjuvant Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-0532
Record Dates: First submitted 2022-11-30; First posted 2022-12-14 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-11

CONDITIONS: Stage I-III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving neoadjuvant therapy

SUMMARY:
In the prospective, open, observational study, we aim to evaluate whether circulating tumor DNA (ctDNA) can be the marker of the response to neoadjuvant therapy in stage I-III breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years-old at the time of consent to participate this trial
* Patients with stage I-III invasive breast cancer
* No prior anti-cancer treatment
* Felt to be a possible candidate for neoadjuvant therapy by their physician

Exclusion Criteria:

* Known to have other aggressive malignant tumor in the past 5 years.
* Breast cancer during lactation; Inflammatory breast cancer; Acute inflammatory disease, pregnancy and other conditions may affect the levels of ctDNA and/or peripheral inflammatory indicators.
* There are other concomitant diseases that seriously threaten the patient's safety or affect the patient's completion of the study, such as serious infection, liver disease, cardiovascular disease, kidney disease, respiratory disease or uncontrolled diabetes or dyslipidemia.
* The investigator determines that subjects are not appropriate to participate in the study due to other factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-III breast cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Miller-Payne grading system | 3 years
Residual cancer burden (RCB) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China